CLINICAL TRIAL: NCT06553989
Title: Impact on Quality of Life of Osteopathic Visceral Mobilizations in Patients Undergoing Post-operative ENDOmetriosis Surgery
Brief Title: Impact on Quality of Life of Osteopathic Visceral Mobilizations After Endometriosis Surgery
Acronym: MOVENDOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RBHP 2023 BOURDEL; 2023-A02653-42 (Other: 2023-A02653-42)
Record Dates: First submitted 2024-08-08; First posted 2024-08-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis; Osteopathy in Diseases Classified Elsewhere
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): patients operated for endometriosis without osteopathic visceral mobilization
- Experimental group (Experimental): patients operated for endometriosis with osteopathic visceral mobilization
  Interventions: Other: osteopatic visceral mobilization

INTERVENTIONS:
Other: osteopatic visceral mobilization — a combination of breathing and visceral mobilizations
  Arms: Experimental group

SUMMARY:
One of the most common post-operative complications of gynaecological surgery, and in particular endometriosis surgery, is the formation of peritoneal adhesions. After laparotomy, it affects up to 90% of patients. Minimally invasive techniques (such as laparoscopy) reduce the risk of adhesion formation, but cannot totally prevent it. Adhesions can lead to chronic pelvic pain, dyspareunia, digestive disorders and infertility. Various strategies and devices have been developed to try and limit adhesion formation, but their effectiveness has not been fully proven in the literature. The only real treatment for adhesions is adhesiolysis, although adhesions often reform. The quality of surgery remains the best means of preventing adhesion formation. To reduce the morbidity associated with pelvic adhesions, it is essential to develop alternative, non-invasive, anti-adhesive methods such as manual osteopathic visceral mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Woman of legal age
* Indication for surgery for infiltrating endometriosis
* Able to give informed consent to participate in research
* Patient included in NO ENDO (national endometriosis observatory promoted by Clermont-Ferrand University Hospital)

Exclusion Criteria:

* Indication for surgery for superficial endometriosis
* Patient of legal age, under guardianship or trusteeship
* Pregnant or breast-feeding patient
* Patients not affiliated to the social security system
* Patients who do not speak French
* Patients under court protection
* Simultaneous participation in another study
* Refusal to participate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life with the EHP-30 questionnaire score | 1 year
  Percentage change in baseline questionnaire score (EHP-30) between pre-operative visit and 1 year.
  The EHP-30 contains 30 items and ranges from 0 (best health) to 100 (worst health). The items in the baseline questionnaire are grouped into 5 main sub-domains: pain, control and powerlessness, emotional well-being, social support and self-image.

SECONDARY OUTCOMES:
quality of life with score of the questionnaire EHP-30 | pre-operative, 6 months and 12 months
  Compare changes in patients' quality of life between the control group and the experimental group with visceral mobilizations
quality of life with score of the questionnaire GIQLI | pre-operative, 6 months and 12 months
  Compare changes in patients' quality of life between the control group and the experimental group with visceral mobilizations
quality of life with score of the questionnaire FSFI | pre-operative, 6 months and 12 months
  Compare changes in patients' quality of life between the control group and the experimental group with visceral mobilizations
quality of life with score of the questionnaire ICIQ-FLUTS | pre-operative, 6 months and 12 months
  Compare changes in patients' quality of life between the control group and the experimental group with visceral mobilizations
quality of life with score of the questionnaire PCS | pre-operative, 6 months and 12 months
  Compare changes in patients' quality of life between the control group and the experimental group with visceral mobilizations
pelvic pain | pre-operative, 6 hours after surgery, 1 day after surgery, 1 month after surgery, 6 months and 12 months
  Compare pelvic pain between the 2 groups using EVA Scale (Visual Analogic Scale (from 0 : no pain to 10 : worst pain possible)
quality of life with the sub-domains of the EHP-30 questionnaire | pre-operative, 6 months and 12 months
  Compare changes in patients' quality of life between the 2 groups regarding the sub-domains the EHP-30 questionnaire
evaluation of the cicatrisation | post operative, 6 months and 12 months
  Examination of scar appearance by the surgeon : acquired healing, healing in progress or disunion
evaluation of the abdominal flexibility | 1 year
  Evaluation of abdominal flexibility with an EVA scale in the regions: right and left iliac fossa, hypogastrium at one year assessed by an independent osteopath between 0 and 10 (0 corresponding to normal flexibility and 10 to total rigidity).
Use of additional care | 1 year
  Compare the use of additional care between the 2 groups by collecting data on the type of consultations (gynecologist, general practitioner, midwife, pain center doctor, emergency doctor, osteopath, physiotherapist, acupuncturist, magnetizer, hypnotherapist, healer, ...) and the number of visits
consumption of analgesics and hormonal treatment | 1 year
  Compare the consumption of analgesics and hormonal treatment (name and dose of the medication) between the 2 groups
fertility | 1 year
  Achieving pregnancy during the first postoperative year (yes or no)
number of days of sick leave | 1 year
  Compare the number of days of sick leave between the two groups
compare patient profiles using the sub-domains of the EHP-30 questionnaire | 1 year
  In the experimental group, identify patient profiles based on the sub-domains of quality of life assessed during the pre-operative visit, and compare these different groups according to the improvement in patients' post-operative quality of life at one year.
patient compliance | 1 year
  evaluate the impact of compliance of patients in the visceral mobilization group on improved quality of life and abdominal flexibility (by collecting the number of osteopathic self-mobilizations performed each month following surgery and during1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bourdel, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France